CLINICAL TRIAL: NCT04915352
Title: Interest of Nasal Provocation Tests for Diagnosis of House Mites Allergic Rhinitis
Acronym: NPT-MAR
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: The study is terminated because the product (nasal provocation test) is out of stock.
Sponsor: Centre Hospitalier Régional Metz-Thionville (Other)
Collaborators: University Hospital, Strasbourg, France (Other); Centre Hospitalier de Verdun (Other); CHU de Reims (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2018-000597-29
Record Dates: First submitted 2021-05-21; First posted 2021-06-07 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Mite Allergy; Respiratory Disease
MeSH Terms: conditions — Respiration Disorders | interventions — Antigens, Dermatophagoides

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Adult dust mite allergenic rhinitis patients (Experimental): Nasal Provocation Test administration (725 Dermatophagoides pteronyssinus (5.000 SBE/ml) dosage form: Lyophilisate and solvent for nasal drops, suspension dosage and frequency: 3 nasal sprays at 3 different concentrations per year: 50, 500 and 5000 SBE / ml for 3 years Duration: 36 months
  Interventions: Drug: Nasal provocation test - 725 Dermatophagoides Pteronyssinus; Other: Negative control

INTERVENTIONS:
Drug: Nasal provocation test - 725 Dermatophagoides Pteronyssinus — 3 different concentrations of Nasal Provocation Test are administered to patients:
  * Nasal spray at 50 SBE/ml for 36 months
  * Nasal spray at 500 SBE/ml for 36 months
  * Nasal spray at 5000 SBE/ml for 36 months
  Other Names: Dermatophagoides Pteronyssinus
Other: Negative control — Negative control using only solvent is applied in order to consider a non-specific nasal hyper reactivity.

SUMMARY:
The aim of this clinical trial is to compare the positive predictive value of the combination rapid nasal provocation test (RNTP) + skin tests (TC) + specific immunoglobulins E (IgEs) to the combination of TC + IgEs (strategy currently used in clinical practice) concerning the efficacy of treatment with Allergen immunotherapy (ITA) at 1 year, in patients with symptoms suggesting allergic rhinitis to house dust mites.

DETAILED DESCRIPTION:
Allergic rhinitis due to house dust mites (AAR) is a common condition which impairs the quality of life of patients and which can be responsible for complications such as the development of asthma. The only curative treatment available is allergenic immunotherapy (ITA).

Currently, the diagnostic approach is based on the history, which collects the symptoms reported by patients during a possible allergen exposure and on the results of skin tests (CT) and / or specific IgE assays (IgEs), which confirm biological sensitization.

In a recent retrospective study, the positive predictive value of TCs and IgEs is estimated at 77% for D. pteronyssinus and 69% for D. farinae. Approximately 30% of patients who have TCs and / or IgEs directed against mites therefore only have biological sensitization.

The nasal challenge test (NPT) has been shown to be an effective tool in improving the diagnosis of dust mite allergic rhinitis. The RNTP is easy to perform, consisting of the nasal spraying of 3 solutions of increasing concentrations (50; 500 and 5000 SBE / ml). RNTP demonstrated good sensitivity and specificity (83.7% and 100%) as well as identical safety in use compared to "classic" TPN. But its real impact on the diagnostic and above all therapeutic strategy has not yet been assessed.

The hypothesis is that RNTP has a positive predictive value superior to TC and IgEs for the diagnosis of allergic rhinitis to dust mites and therefore for the efficacy of ITA.

To demonstrate this, the investigators propose to compare the diagnostic values of these 3 tests, taking the efficacy of ITA at 1 year as the gold standard. The expected results are better predictive values for RNTP, and therefore the possibility of avoiding unnecessary treatments for the patients concerned. About 30% of patients could be treated wrongly now, with the use of TCs and IgEs alone.

ELIGIBILITY:
Inclusion Criteria:

* Patient over 18 years old,
* Patient with persistent mild to severe or moderate to severe intermittent rhinitis according to ARIA criteria, suspicion of allergic rhinitis to dust mites, and a positive skin test for mites and / or a positive mite specific IgE assay
* Patient having signed a free and informed consent

Exclusion Criteria:

* Pregnant or breastfeeding women
* Patients under guardianship or curatorship
* Patients under legal protection
* Patients not affiliated to a social security scheme
* Contraindications to performing a RNPT
* Active ENT or respiratory infections.
* Allergy in acute phase
* History of anaphylaxis due to the allergen involved.
* Unstabilized asthma and other obstructive pathologies.
* Severe general illnesses in evolution.
* Hypersensitivity to one of the components of the product
* Simultaneous treatment with beta-blockers or angiotensin-converting enzyme (ACE) inhibitors,
* Presence of an excessive degree of sensitization (e.g. history, excessive skin reactions),
* Contraindications to immunotherapy:
* Asthma (uncontrolled) or severe [FEV < 70% of the theorical value (after appropriate drug treatment) at the beginning of the treatment].
* Severe asthma exacerbation in the last 3 months
* Active autoimmune diseases
* Malignant tumors
* Pregnancy (initiation of venereal disease)
* AIDS
* Treatment with beta-blockers, including eye drops

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2022-03-07 (Actual); Primary Completion 2024-07-05 (Actual); Study Completion 2024-07-05 (Actual)

PRIMARY OUTCOMES:
The negative predictive value calculated with the efficacy of ITA at 1 year | Year 1
  The primary endpoint is negative predictive value, calculated with the efficacy of ITA at 1 year as the gold standard. It corresponds to the number of patients for whom treatment with an ITA will have been effective at 1 year, divided by the number of patients who have received an ITA.
  It will be calculated on the one hand for patients with TC and / or IgEs positive (control strategy), and on the other hand for patients with TC and / or IgEs positive and RNTP positive.

SECONDARY OUTCOMES:
Efficacity of ITA at 2 and 3 years, according to the same methods as for the primary endpoint. | Years 2 and 3
  The efficacity of ITA at 2nd and 3rd year corresponds to the number of patients for whom treatment with an ITA will have been effective, divided by the number of patients who have received an ITA.
  It will be calculated on the one hand for patients with TC and / or IgEs positive (control strategy), and on the other hand for patients with TC and / or IgEs positive and RNTP positive.
Negative predictive value of the TC + IgEs + RNTP strategy for the efficacy of ITA at 1, 2 and 3 years, according to the same methods as for the primary endpoint. | Years 1, 2 and 3
  The negative predictive value of ITA at 2nd and 3rd year corresponds to the number of patients for whom treatment with an ITA will have been effective, divided by the number of patients who have received an ITA.
  It will be calculated on the one hand for patients with TC and / or IgEs positive (control strategy), and on the other hand for patients with TC and / or IgEs positive and RNTP positive.
Evaluation of the symptoms of allergic rhinitis using the CSMS score at 1, 2 and 3 years | Years 1, 2 and 3
  cSMS: Combined Symptom and Medication Score The European Academy of Allergy and Clinical Immunology published a consensus related to the combination of symptom and medication scores (MSs). The total daily medication score (dMS) ranges from 0 to 3. The CSMS is the sum of total daily symptom score (dSS:range 0-3) and total daily medication score (dMS: range 0-3). Therefore, the values of CSMS are in the range of 0-6 (minmum-maximum).
Assessment of symptoms of allergic rhinitis using Lebel score at 1, 2 and 3 years | Years 1, 2 and 3
  Lebel Bousquet score The RNTP was positive if the (Lebel Bousquet score) was greater than 5/13 points, 13/13 being the worse score
Evaluation of the specific quality of life at 1, 2 and 3 years, using the RQLQ questionnaire. | Years 1, 2 and 3
  Rhinoconjunctivitis Quality of Life Questionnaire (RQLQ) The RQLQ is a self-administered questionnaire that contains 28 questions in 7 domains: activities limitation (3 questions), sleep problems (3 questions), nose symptoms (4 questions), eye symptoms (4 questions), non-nose or eye symptoms (7 questions), practical problems (3 questions), and emotional function (4 questions). Scores for each question range from 0 (not troubled/none of the time) to 6 (extremely troubled/all of the time). The overall RQLQ score is the mean of all 28 responses, and the individual domain scores are the means of the questions in each domain - both range from 0 to 6.

CONTACTS AND LOCATIONS:
Overall Officials: Sébastien LEFEVRE, MD, Principal Investigator — CHR Metz Thionville Hopital de Mercy
Locations (1):
- CHR Metz Thionville/Hopital de Mercy, Metz, Grand Est, France

IPD SHARING:
Plan to Share IPD: No